CLINICAL TRIAL: NCT05201664
Title: Surgical Extrusion: Volumetric and Insertion Analysis at 6 Months. Series of 10 Cases
Brief Title: Surgical Extrusion: Volumetric and Insertion Analysis at 6 Months.
Status: Recruiting | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, DDS, Aula Dental Avanzada
Other Study IDs: EXTQX
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Tooth Extruded; Tooth Extrusion; Tooth Avulsion; Tooth Fracture
Keywords: surgical extrusion; oral surgery; tooth extrusion
MeSH Terms: conditions — Tooth Avulsion; Tooth Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Extrusion: Patients who receive surgical extrusion treatment in maxillary premolars.
  Interventions: Procedure: Surgical Extrusion

INTERVENTIONS:
Procedure: Surgical Extrusion — Relocation of the remaining tooth structure to a more coronal position within the same original socket.

SUMMARY:
The aim is to clinically evaluate the changes that occur in teeth that have undergone surgical extrusion treatment. Three parameters will be recorded before and 6 months after treatment: the position and the volume of the soft tissue, and the level of periodontal attachment.

DETAILED DESCRIPTION:
After informing the patient and obtaining his or her consent to surgical extrusion treatment, a model of the pre-treatment situation will be obtained by intraoral scanning and the attachment levels will be recorded by periodontal probing at 6 points around the tooth.

The dimensional and positional changes of the soft tissue will be analyzed by superimposing both digital impressions in each patient.

In the same way, periodontal attachment levels before and 6 months after treatment will be compared.

The data will be analyzed statistically and conclusions will be drawn regarding the surgical extrusion treatment.

ELIGIBILITY:
Inclusion Criteria:

* Tooth with a subgingival residual dentine margin.
* Patients refusing tooth extraction and dental implant placement as first choice.

Exclusion Criteria:

* Patients in whom surgical intervention is contraindicated.
* Teeth with vertical fractures up to the apex.
* Teeth with pocket depth >4 mm in any of their walls.
* Failure of the treatment leading to the loss of the extruded tooth.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Everyone who attends Clínica Dental Esteve, a private dental clinic in the centre of Alicante.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The position of the soft tissue | 6 months
  Measurement of the vertical position of the gingival margin before and 6 months after surgery.
The volume changes in the soft tissue | 6 months
  Measurement of vestibular alveolar volume before and 6 months after surgery.
The level of insertion | 6 months
  Measurement of the periodontal sulcus before and 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Dental esteve, Alicante, Spain

REFERENCES:
- [Background] Juloski J, Radovic I, Goracci C, Vulicevic ZR, Ferrari M. Ferrule effect: a literature review. J Endod. 2012 Jan;38(1):11-9. doi: 10.1016/j.joen.2011.09.024. Epub 2011 Nov 13. PMID 22152612
- [Background] Khasnis SA, Kidiyoor KH, Patil AB, Kenganal SB. Vertical root fractures and their management. J Conserv Dent. 2014 Mar;17(2):103-10. doi: 10.4103/0972-0707.128034. PMID 24778502
- [Background] Dablanca-Blanco AB, Blanco-Carrion J, Martin-Biedma B, Varela-Patino P, Bello-Castro A, Castelo-Baz P. Management of large class II lesions in molars: how to restore and when to perform surgical crown lengthening? Restor Dent Endod. 2017 Aug;42(3):240-252. doi: 10.5395/rde.2017.42.3.240. Epub 2017 Aug 3. PMID 28808641
- [Background] Bourguignon C, Cohenca N, Lauridsen E, Flores MT, O'Connell AC, Day PF, Tsilingaridis G, Abbott PV, Fouad AF, Hicks L, Andreasen JO, Cehreli ZC, Harlamb S, Kahler B, Oginni A, Semper M, Levin L. International Association of Dental Traumatology guidelines for the management of traumatic dental injuries: 1. Fractures and luxations. Dent Traumatol. 2020 Aug;36(4):314-330. doi: 10.1111/edt.12578. Epub 2020 Jul 17. PMID 32475015
- [Background] Pilalas I, Tsalikis L, Tatakis DN. Pre-restorative crown lengthening surgery outcomes: a systematic review. J Clin Periodontol. 2016 Dec;43(12):1094-1108. doi: 10.1111/jcpe.12617. Epub 2016 Oct 25. PMID 27535216
- [Background] Faria LP, Almeida MM, Amaral MF, Pellizzer EP, Okamoto R, Mendonca MR. Orthodontic Extrusion as Treatment Option for Crown-Root Fracture: Literature Review with Systematic Criteria. J Contemp Dent Pract. 2015 Sep 1;16(9):758-62. doi: 10.5005/jp-journals-10024-1753. PMID 26522603
- [Background] Plotino G, Abella Sans F, Duggal MS, Grande NM, Krastl G, Nagendrababu V, Gambarini G. European Society of Endodontology position statement: Surgical extrusion, intentional replantation and tooth autotransplantation: European Society of Endodontology developed by. Int Endod J. 2021 May;54(5):655-659. doi: 10.1111/iej.13456. Epub 2021 Jan 26. PMID 33501680
- [Background] Gonzalez-Martin O, Carbajo G, Rodrigo M, Montero E, Sanz M. One- versus two-stage crown lengthening surgical procedure for aesthetic restorative purposes: A randomized controlled trial. J Clin Periodontol. 2020 Dec;47(12):1511-1521. doi: 10.1111/jcpe.13375. Epub 2020 Oct 20. PMID 32997836
- [Background] Cordaro M, Staderini E, Torsello F, Grande NM, Turchi M, Cordaro M. Orthodontic Extrusion vs. Surgical Extrusion to Rehabilitate Severely Damaged Teeth: A Literature Review. Int J Environ Res Public Health. 2021 Sep 10;18(18):9530. doi: 10.3390/ijerph18189530. PMID 34574454
- [Background] Das B, Muthu MS. Surgical extrusion as a treatment option for crown-root fracture in permanent anterior teeth: a systematic review. Dent Traumatol. 2013 Dec;29(6):423-31. doi: 10.1111/edt.12054. Epub 2013 Jun 26. PMID 23802693
- [Background] Wang L, Jiang H, Bai Y, Luo Q, Wu H, Liu H. Clinical outcomes after intentional replantation of permanent teeth: A systematic review. Bosn J Basic Med Sci. 2020 Feb 5;20(1):13-20. doi: 10.17305/bjbms.2019.3937. PMID 30684952
- [Background] Mohamed M, Moheb D, Waly N, Abdalsamad A, Elkhadem A. Effects of different splinting times on surgically extruded teeth with a crown-root fracture: A randomized controlled trial. Dent Traumatol. 2021 Apr;37(2):264-274. doi: 10.1111/edt.12624. Epub 2020 Dec 4. PMID 33179388